CLINICAL TRIAL: NCT04186780
Title: Effects of Lentinula Edodes Bar on Lipid Profile and Antioxidant Status in Borderline High Cholesterol Individuals: a Double Blind Randomized Clinical Trial
Brief Title: Effects of Lentinula Edodes Bars on Dyslipidemia and Oxidative Stress in Cholesterol Individuals: Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sorocaba (Other)
Responsible Party: Principal Investigator, Luciane Cruz Lopes, Responsible researcher, University of Sorocaba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 83741818.5.0000.5500
Record Dates: First submitted 2019-11-26; First posted 2019-12-05 (Actual); Results first posted 2020-09-03 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Dyslipidemias
Keywords: Lentinula edodes; Clinical study; Cholesterolemia; Nutraceuticals
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double blind and placebo-controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will not be informed to which group they belong, intervention or control. Who will do the randomization will not be blind, because during treatment she will know which group is eating the bars with Shiitake. The researcher responsible for the pre- and post-treatment evaluation will be blind and will not know the research intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group: patients with borderline cholesterol consumed two cereal bars with Shiitake per day for 66 days.
  Interventions: Other: Shiitake cereal bar
- Placebo group (Placebo Comparator): Patients with borderline cholesterol consumed two placebo cereal bars for 66 days.
  Interventions: Other: Shiitake cereal bar

INTERVENTIONS:
Other: Shiitake cereal bar — patients with borderline cholesterol exposed to bars with Shiitake

SUMMARY:
The daily change in population routine has stimulated the development of health beneficial value added products. Lentinula edodes (Shiitake) is a mushroom with high protein concentration, low lipid content, rich in fiber, minerals, vitamins, antioxidant compounds, β-glucans and chitosan. This is clinical study phase II, randomized, double-blind for analyze in the effect of eating Shiitake bars on cholesterolemia and oxidative stress levels in individuals with borderline cholesterol. Individuals with at least one of the following biochemical markers (total cholesterol, LDL or triglycerides) at the borderline level were recruited through online questionnaire. Individuals (n = 68) were randomly allocated to two groups (Group I - Shiitake free bar (n = 32); Group II - Shiitake bar (n = 36). Each individual underwent blood collection at 0, 33 and 66 days, and received an unidentified opaque bag containing the bars.Biochemical analyzes (triglycerides, total cholesterol, LDL, HDL and glucose) and oxidative stress markers (Catalase, GSH and TBARS) were performed on samples of individuals.

DETAILED DESCRIPTION:
Study design The primary outcome of the study was cholesterolemia, as assessed by total cholesterol levels, triglycerides or low-density lipoproteins (LDL) and high-density lipoproteins (HDL). The secondary outcomes included blood glucose, Body Mass Index (BMI) and oxidative stress biomarkers.

A prospective Phase II, randomized, double blind and placebo-controlled trial was conducted from September 2018 to December 2018. The study accomplished at University of Sorocaba (UNISO), São Paulo State, Brazil. The study was approved (Annex D) by Human Research Ethics Committee from University of Sorocaba (protocol number 2.824.297), in accordance with Resolution 466/2012 of the National Health Council (BRASIL, 2012) and Research Ethics Review Committee (ERC) (WHO, 2016).

Recruitment of individuals For the recruitment of individuals, the disclosure was initiated five months before the start of Phase II trial. The research was published on the website of the University of Sorocaba (UNISO), on social media and folders distributed throughout campus containing a brief explanation about the research, inclusion and exclusion criteria, and contact of the researcher. According to the Resolution 1.170, from Anvisa (National Health Surveillance Agency), Phase II studies are not allowed with less than 12 people; however, the Agency suggests using a minimum of 24 volunteers.

Eligibility Criteria A total of 165 individuals completed the Google online survey.

* Inclusion Criteria Individuals aged from 20 to 65 years old, of both gender, who had at least one of the following biochemical markers at the borderline level (total cholesterol 180 to 239 mg/dL; LDL 130 to 159 mg/dL; triglycerides of 150 to 200 mg/dL), were recruited, diagnosed by biochemical exams with dates recent to the day of recruitment. The be tolerant to bars ingredients and to Shiitake. Availability to attend the date and time of blood collection.
* Exclusion Criteria However, some of them had diseases such as cancer, heart disease, neurodegenerative disease, diabetes, among others. These diseases could be considered as confounders of the study and some recruited people had to be excluded. Pregnant, lactating or hormone replacement women could not participate either.

Individuals were instructed to no change their eating habits and patterns, physical activity level or oral contraceptive use during the study, thus identifying only the effects of Shiitake added to the diet for each individual on the exposed group.

Study Interventions. The study officially started with 68 individuals, who signed an informed term of consent. In the first (Time 0 - T0), in the second (Time 33 days - T33) and in the third (Time 66 days - T66) meetings, the subjects were submitted to nutritional assessment and anamnesis, 24-hour recall of eating habits and eating frequency.

In the first month of the study 4,100 placebo or mushroom bars were produced and in the second month the production was 3,500 bars. According to the Grotto and collaborators (2015), conducted a study evaluating different Shiitake concentrations (100, 400 and 800 mg/Kg/day) to determine the degree of toxicity in animals. Shiitake concentration of 100 mg/Kg/day has been shown to be safe. Besides, the Shiitake sweet bar formulation was approved in the sensory analysis and purchase intention in the previous study.

Randomization The individuals (68) were randomly allocated (using a table of random numbers) into 2 groups: I - Placebo group (n = 32) and II - Intervention group (n = 36). To ensure the daily recommended intake of Shiitake of 100 mg/Kg/day, each participant was weighted to determine the number of bars consumed per day.

The Individuals after nutritional assessment and blood collection, received an unidentified opaque and sealed packed containing individually vacuum bars for a period of T33 days. The patients and the data collector were blind. The bars of the intervention and placebo groups were similar in texture, flavor, aroma and appearance.

After one month, all individuals returned to the University of Sorocaba for new nutritional assessments, receiving more food bars and blood collection with the same double-blind care (T33). At the end of sixty-six days (T66), subjects returned for the last blood collection and final nutritional assessment.

Biochemical Analysis Total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides and glucose were analyzed by commercial kits, following the manufacturer's specifications, in the automated equipment COBAS C111 (Roche®) according to the methodologies below.

For cholesterol, 10 µL of sample and 1.0 mL of enzyme reagent were mixed at 37 ºC for 10 min for total transformation into free cholesterol, by lipoprotein lipase enzyme. The reaction involved the oxidation of free cholesterol to cholesterol-3-one and H2O2 by the cholesterol oxidase enzyme. And with the action of peroxidase on phenol with 4-aminoantipyrine formed a cherry chromogen, the color being proportional to the concentration of cholesterol.

For the determination of HDL, the serum was treated with phosphotungstate acid and magnesium chloride. So, the LDL was precipitated out from the fraction after centrifugation for 2 min at 10.000 rpm. HDL, which remained in the supernatant, was performed according to the cholesterol methodology. HDL concentration is proportional to the color. LDL was calculated by subtracting HDL cholesterol from total cholesterol.

Serum triglycerides were hydrolyzed to glycerol and free fatty acid by lipoprotein lipase. In the presence of adenosine triphosphate (ATP) and glycerol kinase, glycerol-3-phosphate was phosphorylated, which was oxidized to acetone dihydrogen phosphate and H2O2 by the glycerol phosphate oxidase. H2O2, 4-aminoantipyrine and p-chlorophenol underwent the same reaction process reported above by peroxidase in a 37 ºC water bath for 10 minutes until formation of red color.

For the blood glucose test, glucose-6-phosphate dehydrogenase oxidized glucose-6-phosphate in the presence of NADP in gluconate-6-phosphate. No other carbohydrates have been oxidized. The rate of NADPH formation during the reaction was directly proportional to the glucose concentration, being determined photometrically.

Oxidative Stress Analysis The determination of reduced glutathione (GSH) was made by quantification of reduced total thiols based. For this, 150 µL of the blood was vortexed with 100 µL 10% Triton X-100 and 100 µL 30% TCA, then centrifuged for 10 min at 4000 rpm. In the cuvette 900 µL of 1M TFK, 50 µL of supernatant, and 50 µL of 10 mM DTNB were pipetted, which reacted to form a yellow complex. The reading was taken at 412 nm in a spectrophotometer. For the calculation of concentration, the calibration curve with predefined GSH concentrations (0.005; 0.01; 0.025; 0.05; 0.1 mM) was used.

To evaluate the activity of the catalase enzyme was used, based on the decomposition of H2O2 by catalase, monitored at 240 nm. For this, the blood was diluted 60 times in 50 mM TFK. An aliquot of 20 μL was mixed to 1910 μL of the same TFK, and 70 μL of H2O2 was added, initiating the monitored reaction for three minutes. A constant of variation (κ) per minute helped in the expression of catalase enzyme (κ/min).

Thiobarbituric acid reactive substances (TBARS) were used as a biomarker of lipid peroxidation. Plasma aliquots (150 µL) were mixed with 50 µL NaOH and 50 µL Milli-Q ultrapure water (Direct 8, Millipore®) and incubated at 60 °C for 30 minutes with shaking. 250 µL of 6% H₃PO₄, 250 µL of 0.8% TBA and 100 µL of 10% SDS were added to the samples and taken to the 80 °C bath for one hour. Lipid peroxides reacted with TBA in acidic medium to form a pink compound and read in a spectrophotometer at 532 nm. To calculate the concentration of TBARS in plasma, a calibration curve of malondialdehyde, the main thiobarbituric acid reactive substance, was made (0.28; 0.56; 1.7; 3.4; 6.6 µM).

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged from 20 to 65 years old, of both gender, who had at least one of the following biochemical markers at the borderline level (total cholesterol 180 to 239 mg/dL; LDL 130 to 159 mg/dL; triglycerides of 150 to 200 mg/dL), were recruited, diagnosed by biochemical exams with dates recent to the day of recruitment. The be tolerant to bars ingredients and to Shiitake. Availability to attend the date and time of blood collection.

Exclusion Criteria:

* However, some of them had diseases such as cancer, heart disease, neurodegenerative disease, diabetes, among others. These diseases could be considered as confounders of the study and some recruited people had to be excluded. Pregnant, lactating or hormone replacement women could not participate either.

Individuals were instructed to no change their eating habits and patterns, physical activity level or oral contraceptive use during the study, thus identifying only the effects of Shiitake added to the diet for each individual on the exposed group

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula M Bertoni, MSc, Study Chair — University of Sorocaba; Miriam SN Silveira, MSc, Study Chair — University of Sorocaba
Locations (1):
- University of Sorocaba, Sorocaba, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
After the article publication will be shared the data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After January 2021
Access Criteria: Anyone can access the information.

REFERENCES:
- [Background] Aebi H. Catalase in vitro. Methods Enzymol. 1984; 105: 121-126. Ellman GL. Tissue sulfhydryl groups. Arch Biochem Biophys. 1959; 82: 70-77. Friedewald, W. T.; LEVY, R. I.; Frederickson, D. S. Estimation of the concentration of low density lipoprotein in plasma without the use of the preparative ultra centrifuge. Clinical Chemistry. 1972; 18(6): 499-502 Grotto D, Gerenutti M, Souza VCO, Barbosa F Jr. Deficiency of macro and micronutrients induced by Lentinula edodes. Toxicology. 2015. 2:401-404.. Kerckhoffs DAJM, Hornstra G, Mensink RP. Cholesterol-lowering effect of β-glucan from oat bran in mildly hypercholesterolemic subjects may decrease when β-glucan is incorporated into bread and cookies. American Journal of Clinical Nutrition. 2003; 78: 221-227. Ohkawa H, OhishI N, Yagi K. Assay for lipid peroxides in animal tissues by Thiobarbituric Acid reaction. Analyt Biochem. 1979; 95: 351-358.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were received in September, October and November in the nursing room at the University for the meetings.
Pre-assignment Details: Individuals aged from 20 to 65 years old, who had at least one of the following biochemical markers at the borderline level, were recruited. Must be tolerant to bars ingredients and to Shiitake and they must be availability to attend the date and time of blood collection.
  Some of the individuals had diseases such as cancer, heart disease, neurodegenerative disease, diabetes, among others. These diseases could be confounders of the study and some recruited people had to be excluded.
Groups:
- Placebo Group: Patients with borderline cholesterol consumed two placebo cereal bars for 66 days.
  Placebo cereal bar: patients with borderline cholesterol exposed to cereal bars without Shiitake.
Period: Overall Study
Arm/Group | Intervention Group | Placebo Group
Started | 36 | 32
Completed | 22 | 25
Not Completed | 14 | 7

BASELINE CHARACTERISTICS:
Population: Analyzed the effects of Shiitake ingestion by supplemented bars on borderline cholesterol and oxidative stress in humans through a phase II, double-blind randomized trial.
Groups:
- Placebo Group: Patients with borderline cholesterol consumed two placebo cereal bars for 66 days.
  Cereal bar: patients with borderline cholesterol exposed to placebo cereal bars.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Placebo Group | Total
Number analyzed (Participants) | 36 | 32 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 32 | 68
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42 (12) | 38 (11) | 40 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 23 | 53
  Male | 6 | 9 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 36 | 32 | 68
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 36 | 32 | 68
Measure Smoker tobacco [Count of Participants; unit: Participants] | 2 | 4 | 6
Number of Participants Reporting Alcohol Consumption [Count of Participants; unit: Participants] | 19 | 14 | 33
Number of Participants Reporting Regular Physical Activity [Count of Participants; unit: Participants] | 14 | 17 | 31
BMI - Body mass index [Mean (Standard Deviation); unit: kg/m²] | 26.4 (4.4) | 27.5 (4.4) | 26.9 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Total Cholesterol Levels
Description: Total cholesterol It was analyzed by commercial kits, according to the manufacturer's specifications. The volunteers' Total Cholesterol and Triglyceride levels were analyzed at Time 0 (when starting the study), at Time 33 (after 33 days) and at Time 66 (after 66 days).
Time Frame: Assessed at 0, 33 and 66 days. Days 0 and 66 reported.
Population: Individuals aged from 20 to 65 years old, of both gender, who had at least one of the following biochemical markers at the borderline high level (total cholesterol 180 to 239 mg/dL; LDL 130 to 159 mg/dL; TG of 150 to 200 mg/dL)
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Placebo Group: Participants received two placebo food bars/day to consume for 66 days. Placebo: Placebo food bars with 25 g each.
- Intervention Group: Participants received two shiitake food bars/day to consume for 66 days. Intervention group: Shiitake bars with 25 g each.
Arm/Group | Placebo Group | Intervention Group
Number analyzed (Participants) | 32 | 36
mg/dL
  Total Cholesterol T0 | 222.8 (33.1) | 228.2 (45.4)
  Total Cholesterol T66 | 226.7 (41.3) | 229.6 (38.2)
Statistical Analysis 1: Comparison: Placebo Group vs Intervention Group; Test type: Superiority — The differences between Shiitake and placebo groups were analyzed by the Chi-square test, Exact of Fisher test and Student's t-test. Descriptions of all biochemical parameters were expressed as mean ± standard deviation. To investigate the differences in biochemical parameters between the groups, Analysis of Variance (ANOVA) with repeated measurements was applied. All results of biochemical parameters were normalized to logarithmic scale; p = 0.59, ANOVA — P < 0.05 was accepted as statistically significant; Mean Difference (Net) = 2.5 — Difference between T0 and T66 in the placebo group and intervention group in total cholesterol

2. Secondary Outcome: Oxidative Stress: Catalase
Description: The activity of the catalase enzyme was based on the decomposition of H2O2, monitored at 240 nm. A constant of variation or coefficient of variation (κ) per minute helped in the expression of catalase enzyme (κ/min). The Catalase enzyme has the responsibility to break down hydrogen peroxide. Higher scores mean a better outcome.
  Were analyzed at Time 0 (when starting the study), at Time 33 (after 33 days) and at Time 66 (after 66 days).
Time Frame: Assessed at 0, 33 and 66 days. Days 0 and 66 reported.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: k/min
Groups:
- Placebo Group: Participants received two placebo bars/day to consume for 66 days. Placebo group: Bars with 25 g each.
- Intervention Group: Participants received two shiitake bars/day to consume for 66 days. Intervention: Shiitake bars with 25 g each.
Arm/Group | Placebo Group | Intervention Group
Number analyzed (Participants) | 32 | 36
k/min
  Catalase T0 | 3.5 (1.1) | 3.1 (0.8)
  Catalase T66 | 3.7 (1.6) | 3.7 (2.0)
Statistical Analysis 1: Comparison: Placebo Group vs Intervention Group; Test type: Superiority — The differences between Shiitake and placebo groups were analyzed by the Chi-square test, Exact of Fisher test and Student's t-test. Descriptions of all biochemical and oxidative stress parameters were expressed as mean ± standard deviation. To investigate the differences in biochemical parameters between the groups, Analysis of Variance (ANOVA) with repeated measurements was applied. All results of biochemical parameters and oxidative stress were normalized to logarithmic scale; p = 0.8284, ANOVA — P < 0.05 was accepted as statistically significant; Mean Difference (Net) = 0.4 — Difference between T0 and T66 in the placebo group and intervention group

3. Secondary Outcome: Oxidative Stress: Reduced Glutathione (GSH)
Description: Reduced Glutathione was analyzed in the volunteers' samples at Time 0 (at the beginning of the study), at Time 33 (after 33 days) and at Time 66 (after 66 days).
Time Frame: Assessed at 0, 33 and 66 days. Days 0 and 66 reported.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | Placebo Group | Intervention Group
Number analyzed (Participants) | 32 | 36
mM
  GSH T0 | 0.4 (0.1) | 0.4 (0.2)
  GSH T66 | 0.6 (0.2) | 0.5 (0.2)
Statistical Analysis 1: Comparison: Placebo Group vs Intervention Group; Test type: Superiority; p = 0.0058, ANOVA — P < 0.05 was accepted as statistically significant; Median Difference (Net) = 0.1 — Difference between T0 and T66 in the placebo group compared to the intervention group

4. Secondary Outcome: Oxidative Stress: Thiobarbituric Acid Reactive Substances (TBARS)
Description: Reactive Substances to Thiobarbituric Acid were analyzed in the volunteers' samples at Time 0 (at the beginning of the study), at Time 33 (after 33 days) and at Time 66 (after 66 days).
Time Frame: Assessed at 0, 33 and 66 days. Days 0 and 66 reported.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Placebo Group | Intervention Group
Number analyzed (Participants) | 32 | 36
µM
  TBARS T0 | 13.9 (2.3) | 14.6 (2.1)
  TBARS T66 | 14.7 (2.0) | 13.9 (2.9)
Statistical Analysis 1: Comparison: Placebo Group vs Intervention Group; Test type: Superiority; p = 0.0384, ANOVA — P < 0.05 was accepted as statistically significant; Median Difference (Net) = 0.8 — Reduced difference in TBARS in the placebo group compared to the intervention group at T66

5. Primary Outcome: Triglycerides Levels
Description: The triglycerides levels It was analyzed by commercial kits, according to the manufacturer's specifications. The volunteers' Total Cholesterol and Triglyceride levels were analyzed at Time 0 (when starting the study), at Time 33 (after 33 days) and at Time 66 (after 66 days).
Time Frame: Assessed at 0, 33 and 66 days. Days 0 and 66 reported.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Group | Intervention Group
Number analyzed (Participants) | 32 | 36
mg/dL
  Triglycerides T0 | 144.5 (70.2) | 178.9 (170.1)
  Triglycerides T66 | 207.7 (202.7) | 160.7 (94.7)
Statistical Analysis 1: Comparison: Placebo Group vs Intervention Group; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0352, ANOVA — P < 0.05 was accepted as statistically significant; Mean Difference (Net) = 47.0 — Difference between placebo group and intervention group of T66

ADVERSE EVENTS:
Time Frame: 15 days
Description: 7 patients communicated the manifestation of the allergic reaction.
Groups:
- Intervention Group: Intervention group: patients with borderline cholesterol consumed two cereal bars with Shiitake per day for 66 days.
  The patients can manifest allergy to ingredients the bars
- Placebo Group: Patients with borderline cholesterol consumed two placebo cereal bars for 66 days.
  The patients can manifest allergy to ingredients the bars.
Arm/Group | Intervention Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/32
Other Adverse Events (participants affected / at risk) | 7/36 | 0/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=36) | Placebo Group (N=32)
Allergic Reaction (Skin and subcutaneous tissue disorders) | 7 (36) | NA (32)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT04186780/SAP_000.pdf
  • Study Protocol (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT04186780/Prot_003.pdf
  • Informed Consent Form (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT04186780/ICF_004.pdf